CLINICAL TRIAL: NCT06886620
Title: A Phase III Prospective, Randomized, Double Blind, Active Controlled, Multicenter, Parallel Group Study to Assess the Safety and Effectiveness of Once Daily PMR Compared to Twice Daily Pletaal® in Patients With Intermittent Claudication
Brief Title: Assess the Safety and Effectiveness of Once Daily PMR Compared to Twice Daily Pletaal® in Patients With Intermittent Claudication
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBL14-001
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Intermittent Claudication
Keywords: Peripheral Arterial Disease; Ankle Brachial Index; Absolute Claudication Distance; Initial Claudication Distance; PMR; Cilostazol
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PMR (Experimental): Cilostazol 200 mg, tablet, PO, QN
  Interventions: Drug: Cilostazol 200 mg
- Pletaal® (Active Comparator): Cilostazol 100 mg, tablet, PO, BID
  Interventions: Drug: Cilostazol 100 mg

INTERVENTIONS:
Drug: Cilostazol 200 mg — Provided as 1# placebo tablet in the morning and 1# PMR 200 mg/tablet in the evening, orally, for 24 weeks.
  Other Names: PMR
  Arms: PMR
Drug: Cilostazol 100 mg — Provided as 1# Pletaal® 100 mg/tablet, orally twice a day, for 24 weeks.
  Other Names: Pletaal®
  Arms: Pletaal®

SUMMARY:
The study is designed to compare the efficacy and safety of once daily PMR treatment with twice daily Pletaal® treatment in patients with intermittent claudication caused by peripheral arterial disease and are currently treated with cilostazol of any strength and any dosing frequency.

ELIGIBILITY:
Main Inclusion Criteria:

* Stable use of Cilostazol of any strength and any dosing frequency for at least 3 months prior to screening, for the treatment of peripheral arterial disease.
* Initial claudication distance ≥ 30 meters at the constant workload treadmill test.

Main Exclusion Criteria:

* Presence of limb-threatening chronic limb ischemia, manifested by ischemic rest pain, ulceration or gangrene.
* History of lower-extremity surgical or endovascular arterial reconstructions or sympathectomy within 3 months prior to screening.
* Presence of illness(es) (such as angina pectoris, respiratory disease, orthopaedic disease, or neurological disorders, except the study disease) limiting the exercise capacity.
* Presence of uncontrolled hypertension (based on physician's judgment) or other unstable cardiovascular disease such as congestive heart failure of any severity and myocardial infarction within 6 months prior to screening.
* History of coronary artery bypass graft (CABG) or major cardiovascular surgical procedures within 6 months prior to screening.
* History of Buerger's disease or deep vein thrombosis within 3 months prior to screening.
* Presence of haemostatic disorders or active pathologic bleeding, such as bleeding peptic ulcer and intracranial bleeding.
* Presence or history of ventricular tachycardia, ventricular fibrillation or multifocal ventricular tachycardia with or without adequate treatment, QTc prolongation associated with cardiac disorders, or severe tachyarrhythmia within 6 months prior to screening, which is considered not suitable for this study by Investigator.
* History of type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus.
* Use of anticoagulant agent(s) within 6 months prior to screening.
* Use of two or more than two anti-platelet agents within 3 months prior to screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Geometric mean percent change in initial claudication distance (ICD) | At baseline (day 0) and week 24
  The standardized workload treadmill test will be conducted for evaluation of walking performance.
  ICD is defined as the distance walked to the point of the onset of claudication symptoms.

SECONDARY OUTCOMES:
Geometric mean percent change in initial claudication distance (ICD) | At baseline (day 0) and week 12
  The standardized workload treadmill test will be conducted for evaluation of walking performance.
  ICD is defined as the distance walked to the point of the onset of claudication symptoms.
Geometric mean percent change in absolute claudication distance (ACD) | At baseline (day 0) and week 12
  The standardized workload treadmill test will be conducted for evaluation of walking performance.
  ACD is defined as the maximal distance walked to the point where severe claudication pain forced cessation of exercise.
Geometric mean percent change in absolute claudication distance (ACD) | At baseline (day 0) and week 24
  The standardized workload treadmill test will be conducted for evaluation of walking performance.
  ACD is defined as the maximal distance walked to the point where severe claudication pain forced cessation of exercise.
Subject assessment of treatment response | At week 24
  Participants will subjectively evaluate the treatment response of study drug on claudication symptoms which will be categorized into:
  * Much Better
  * Better
  * Unchanged
  * Worse
  * Much Worse
  Participants rating their improvement on claudication symptoms as "Much Better" or "Better" are classified as responders.

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Kuang Lee, M.D., Principal Investigator — National Taiwan University Hospital; Chern-En Chiang, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan; Jen-Yuan Kuo, M.D., Principal Investigator — Mackay Memorail Hospital; Ming-Shien Wen, M.D., Principal Investigator — Chang Gung Memorial Hospital; Yin-Wei Hsian, M.D., Ph.D., Principal Investigator — Cheng-Hsin General Hospital
Locations (5):
- Taiwan (5):
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No